CLINICAL TRIAL: NCT06865768
Title: Prospective Phase II Validation of the Performance of a Prostate-Specific Membrane Antigen (PSMA) Radiotracer for Positron Emission Tomography-Multiparametric Magnetic Resonance (PET-mpMR) Imaging to Target Prostate Biopsy Via Transrectal Ultrasound (TRUS) -Magnetic Resonance Imaging (MRI) Fusion Technique
Brief Title: An Investigational Scan (18F-rhPSMA-7.3 PET-mpMRI) for Targeted Prostate Biopsy Using TRUS-MR Fusion Technique
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David M Schuster, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00007915; NCI-2025-00207 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00007915 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6265-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH); U01CA113913 (NIH)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Masking Description: MR interpreters will be blinded to PET findings
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (18F-rhPSMA-7.3 PET, mpMRI, TRUS-MR fusion biopsy) (Experimental): Patients receive 18F-rhPSMA-7.3 IV and, 50 minutes later, undergo PET over 30 minutes at the time of SOC mpMRI. Patients may also undergo standard of care TRUS-MR fusion biopsy of targets identified on SOC mpMRI.
  Interventions: Drug: Flotufolastat F-18 Gallium; Procedure: Magnetic Resonance Imaging; Procedure: Multiparametric Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Transrectal Ultrasonography Guided Biopsy

INTERVENTIONS:
Drug: Flotufolastat F-18 Gallium — Given IV
  Other Names: (18F)-rhPSMA-7.3; 18F-rhPSMA-7.3; 18FrhPSMA-7.3; F-18-rhPSMA-7.3; Fluorine F 18 Radiohybrid PSMA-7.3; Fluorine F 18 rhPSMA-7.3; Fluorine-18 rhPSMA-7.3; Posluma; rhPSMA-7.3 (18F)
Procedure: Magnetic Resonance Imaging — Undergo TRUS-MR fusion biopsy
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo mpMRI
  Other Names: MP-MRI; mpMRI; Multi-parametric MRI; Multiparametric MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Transrectal Ultrasonography Guided Biopsy — Undergo TRUS-MR fusion biopsy
  Other Names: TRUS Biopsy; TRUS-Guided Biopsy

SUMMARY:
This phase II trial evaluates an imaging technique called 18F-rhPSMA-7.3 positron emission tomography (PET)-multiparametric (mp) magnetic resonance imaging (MRI) in identifying tumor tissue in men suspected to have prostate cancer. This clinical trial also seeks to determine if the abnormal tissue identified during imaging represents the tumor tissue removed during transrectal ultrasound-magnetic resonance imaging (TRUS-MR) fusion biopsy of the prostate. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of tracer, in the case of this research, 18F-rhPSMA-7.3. Because some tumors take up 18F-rhPSMA-7.3 it can be seen with PET. MRI uses radio waves and a powerful magnet linked to a computer to create detailed pictures of areas inside the body. These pictures can show the difference between normal and diseased tissue. Standard of care imaging for prostate cancer includes mpMRI, which is the combination of multiple magnetic resonance techniques, including diffusion weighted imaging, dynamic contrast-enhanced imaging, and spectroscopy, to achieve an image that will allow for better identification of tumor size and location, as well as possibly identifying tumor spread and aggressiveness. However, mpMRI may not be as effective in identifying prostate tumors that are clinically significant. A TRUS-MR biopsy involves using both ultrasound and MRI scans to locate abnormal areas in the prostate. An 18F-rhPSMA-7.3 PET-mpMRI may be more effective than mpMRI alone in identifying tumor tissue and may increase the accuracy of TRUS-MRI fusion biopsies in men suspected of having prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if simultaneous flotufolastat F-18 gallium (18F-rhPSMA-7.3) PET-mpMR improves the detection of clinically significant prostate cancer (csPCa) in Prostate Imaging-Reporting and Data System (PI-RADS) ≥ 3 lesions.

SECONDARY OBJECTIVE:

I. To explore associations between radiomics textural data from the PET acquisition, mpMR imaging, or both with the presence of csPCa.

OUTLINE:

Patients receive 18F-rhPSMA-7.3 intravenously (IV) and, 50 minutes later, undergo PET over 30 minutes at the time of standard of care (SOC) mpMRI. Patients may also undergo standard of care TRUS-MR fusion biopsy of targets identified on SOC mpMRI.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged > 18 years
* Patients with suspected prostate cancer who will have prostate biopsy for confirmation
* Ability to lie still for MRI scanning
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Documented acute prostatitis, symptomatic or severe benign prostatic hyperplasia (BPH) or urinary tract infections
* Patients with contraindications for MRI including implantable pace makers, cochlear implants
* Patients with uni- or bilateral hip prosthesis
* Subjects with other significant medical conditions that would create unacceptable prostate biopsy risk, compromise retention on study or compromise study related assessments
* Prostate biopsy within 4 weeks prior to entry on this study in which inflammation might affect PET-mpMR result
* Is determined by the Investigator that the patient is clinically unsuitable for the study
* Is incapable of understanding the language in which the information for the patient is given
* Participation in a concurrent clinical trial or in another trial within the past 30 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Discrimination of clinically significant prostate cancer (csPCa) from non-csPCa | Up to 3 months from imaging scan
  Will determine if radiotracer activity within the sampled regions improves discrimination of csPCa from non-csPCa. The receiver operating characteristic and its associated area under the curve (AUC) for positron emission tomography standardized uptake value maximum will be estimated. To accommodate within-individual correlation among multiple lesions, 95% confidence intervals for the AUC will be obtained through bootstrap with re-sampling of patients.

CONTACTS AND LOCATIONS:
Overall Officials: David M Schuster, MD, FACR, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States